CLINICAL TRIAL: NCT00003052
Title: Randomized Study Comparing Neoadjuvant Chemotherapy Etoposide + Ifosfamide + Adriamycin (EIA) Combined With Regional Hyperthermia (RHT) Versus Neoadjuvant Chemotherapy Alone in the Treatment of High-Risk Soft Tissue Sarcomas in Adults
Brief Title: Combination Chemotherapy With or Without Hyperthermia Therapy in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: The European Society for Hyperthermic Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065699; EORTC-62961
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-11

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; adult extraskeletal osteosarcoma; adult malignant fibrous histiocytoma; adult rhabdomyosarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Rhabdomyosarcoma | interventions — Doxorubicin; Etoposide; Ifosfamide; Diathermy; Radiotherapy

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Procedure: conventional surgery
Procedure: hyperthermia treatment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. It is not known whether receiving chemotherapy plus hyperthermia is more effective than receiving chemotherapy alone in treating patients with soft tissue sarcoma.

PURPOSE: This randomized phase III trial is studying combination chemotherapy alone to see how well it works compared to combination chemotherapy and hyperthermia therapy in treating patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine local progression-free survival of patients with high-risk soft tissue sarcoma treated with neoadjuvant etoposide, ifosfamide, and doxorubicin with or without regional hyperthermia.
* Determine the tumor response rate, local disease control rate, and overall survival in patients treated with this regimen.

OUTLINE: This is a randomized study. Patients are stratified according to high-risk category (S1 vs S2 vs S3) and disease site (extremity vs nonextremity). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive etoposide IV over 30 minutes on days 1 and 4, ifosfamide IV over 60 minutes on days 1-4, and doxorubicin IV over 30 minutes on day 1. Treatment continues every 21 days for a total of 4 courses. Patients also undergo regional hyperthermia.
* Arm II: Patients receive chemotherapy alone as in arm I. Patients in both arms undergo definitive surgery 4-6 weeks after chemotherapy. Patients also undergo radiotherapy beginning 4-6 weeks after surgery. After completion of surgery and radiotherapy, patients with non-resectable tumors showing no disease progression receive an additional 4 courses of chemotherapy with or without regional hyperthermia according to above treatment schedule.

Patients are followed every 3 months for 1 year, every 4 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 340 patients (170 patients per arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven grade II or III soft tissue sarcoma of one of following high-risk groups:

  * Grade II/III primary tumor with lesion size of at least 5 cm, deep, and extracompartmental (S1)
  * Local recurrence of primary tumor (S2)
  * Inadequate surgical excision of S1 or S2 (S3)
* Disease recurrence after prior surgery allowed
* The following histological types are eligible:

  * Malignant fibrous histiocytoma
  * Liposarcoma (round cell and pleomorphic)
  * Leiomyosarcoma
  * Fibrosarcoma
  * Rhabdomyosarcoma
  * Synovial sarcoma
  * Malignant paraganglioma
  * Neurofibrosarcoma (malignant schwannoma)
  * Extraskeletal Ewing's sarcoma
  * Extraskeletal osteosarcoma
  * Malignant peripheral neuroectodermal tumors
  * Mesenchymal chondrosarcoma
  * Angiosarcoma
  * Miscellaneous sarcoma
  * Unclassified sarcoma
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* WHO 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding disorder

Hepatic:

* Bilirubin less than 1.25 times upper limit of normal
* No severe hepatic dysfunction

Renal:

* Creatinine clearance greater than 60 mL/min
* No chronic renal failure

Cardiovascular:

* No documented existing cardiac failure
* No manifest heart failure (New York Heart Association class III or IV)
* Left ventricular ejection fraction no more than 10% below institutional normal

Other:

* No other prior or concurrent malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No other severe disease
* No severe cerebrovascular disease
* No extremely obese patients
* No prior metallic implants relevant to the regional hyperthermia field
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy (except to disease recurrence outside study irradiation field)

Surgery:

* See Disease Characteristics
* No prior mutilative surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 1997-07; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Local progression-free survival

SECONDARY OUTCOMES:
Response as assessed by WHO criteria
Overall survival
Relapse-free survival
Acute and late complications as assessed by CTC v 1.0

CONTACTS AND LOCATIONS:
Overall Officials: Rolf D. Issels, MD, PhD — Klinikum der Universitaet Muenchen - Grosshadern Campus; Rolf D. Issels, MD, PhD, Study Chair — Klinikum der Universitaet Muenchen - Grosshadern Campus
Locations (4):
- Germany (4):
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich

REFERENCES:
- [Background] Stahl R, Wang T, Lindner LH, Abdel-Rahman S, Santl M, Reiser MF, Issels RD. Comparison of radiological and pathohistological response to neoadjuvant chemotherapy combined with regional hyperthermia (RHT) and study of response dependence on the applied thermal parameters in patients with soft tissue sarcomas (STS). Int J Hyperthermia. 2009 Jun;25(4):289-98. doi: 10.1080/02656730902873616. PMID 19670096
- [Result] Issels RD, Lindner LH, Verweij J, Wust P, Reichardt P, Schem BC, Abdel-Rahman S, Daugaard S, Salat C, Wendtner CM, Vujaskovic Z, Wessalowski R, Jauch KW, Durr HR, Ploner F, Baur-Melnyk A, Mansmann U, Hiddemann W, Blay JY, Hohenberger P; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group (EORTC-STBSG); European Society for Hyperthermic Oncology (ESHO). Neo-adjuvant chemotherapy alone or with regional hyperthermia for localised high-risk soft-tissue sarcoma: a randomised phase 3 multicentre study. Lancet Oncol. 2010 Jun;11(6):561-70. doi: 10.1016/S1470-2045(10)70071-1. Epub 2010 Apr 29. PMID 20434400
- [Result] Issels RD, Lindner LH, Wust P, et al.: Regional hyperthermia (RHT) improves response and survival when combined with systemic chemotherapy in the management of locally advanced, high grade soft tissue sarcomas (STS) of the extremities, the body wall and the abdomen: a phase III randomised pros. [Abstract] J Clin Oncol 25 (Suppl 18): A-10009, 547s, 2007.
- [Result] Lindner LH, Schlemmer M, Hohenberger P, et al.: Risk assessment of early progression among 213 pts with high-risk soft tissue sarcomas (HR-STS) treated with neoadjuvant chemotherapy regional hyperthermia: EORTC 62961/ESHO-RHT 95 intergroup phase III study. [Abstract] J Clin Oncol 23 (Suppl 16): A-9020, 821s, 2005.
- [Derived] Issels RD, Noessner E, Lindner LH, Schmidt M, Albertsmeier M, Blay JY, Stutz E, Xu Y, Buecklein V, Altendorf-Hofmann A, Abdel-Rahman S, Mansmann U, von Bergwelt-Baildon M, Knoesel T. Immune infiltrates in patients with localised high-risk soft tissue sarcoma treated with neoadjuvant chemotherapy without or with regional hyperthermia: A translational research program of the EORTC 62961-ESHO 95 randomised clinical trial. Eur J Cancer. 2021 Nov;158:123-132. doi: 10.1016/j.ejca.2021.09.015. Epub 2021 Oct 16. PMID 34666214
- [Derived] Issels RD, Lindner LH, Verweij J, Wessalowski R, Reichardt P, Wust P, Ghadjar P, Hohenberger P, Angele M, Salat C, Vujaskovic Z, Daugaard S, Mella O, Mansmann U, Durr HR, Knosel T, Abdel-Rahman S, Schmidt M, Hiddemann W, Jauch KW, Belka C, Gronchi A; European Organization for the Research and Treatment of Cancer-Soft Tissue and Bone Sarcoma Group and the European Society for Hyperthermic Oncology. Effect of Neoadjuvant Chemotherapy Plus Regional Hyperthermia on Long-term Outcomes Among Patients With Localized High-Risk Soft Tissue Sarcoma: The EORTC 62961-ESHO 95 Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):483-492. doi: 10.1001/jamaoncol.2017.4996. PMID 29450452
- [Derived] Knosel T, Altendorf-Hofmann A, Lindner L, Issels R, Hermeking H, Schuebbe G, Gibis S, Siemens H, Kampmann E, Kirchner T. Loss of p16(INK4a) is associated with reduced patient survival in soft tissue tumours, and indicates a senescence barrier. J Clin Pathol. 2014 Jul;67(7):592-8. doi: 10.1136/jclinpath-2013-202106. Epub 2014 Apr 19. PMID 24747207